CLINICAL TRIAL: NCT02000739
Title: Phase II GENIUS Trial of GENetically-Informed Therapies for Patients With previoUSly Treated Refractory Metastatic Cancer
Brief Title: Genetically-informed Therapies for Patients With Metastatic Cancer
Acronym: GENIUS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D13214
Record Dates: First submitted 2013-11-06; First posted 2013-12-04 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Metastatic Cancer
Keywords: Breast cancer; melanoma; GI cancer; ovarian cancer; lung cancer; metastatic cancer; brain cancer; head and neck cancer
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Melanoma; Gastrointestinal Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Brain Neoplasms; Head and Neck Neoplasms | interventions — Patient-Specific Modeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genetically Informed Therapy (Other): The treatment participants get will depend on the results of the DNA sequencing and the availability of targeted therapies that match the genetic profile of the tumor identified by the DNA sequencing.
  If there is a genetic mutation that can be identified with current DNA sequencing and a drug has been developed for this mutation, participants may be able to receive that drug. If there is more than one drug available, the participant and his/her oncologist will decide which is the best one for the participant.
  Interventions: Genetic: Genetically Informed Therapy

INTERVENTIONS:
Genetic: Genetically Informed Therapy — If there is a genetic mutation that can be identified with current DNA sequencing and a drug has been developed for this mutation, participants may be able to receive that drug. If there is more than one drug available, the participant and his/her oncologist will decide which is the best one for the participant.
  Other Names: Patient Specific

SUMMARY:
Genetic mutations associated with cancer are being discovered and new treatments are being created to treat people whose cancer tumors have certain genetic mutations. Genetic sequencing of a tumor can be done, and in this study that information is sent to a company called "N-of-One." They will match each patient's tumor's genetic profile to targeted therapies. The targeted therapies may be use of FDA-approved drugs, off-label use of FDA-approved drugs, or use of experimental drugs in clinical research studies open at various locations in the region.

The purpose of the study is to compare the length of time it takes for a tumor to grow in people who receive the standard treatment for metastatic cancer to the length of time it takes for a tumor to grow in people who receive a drug specifically targeted for their cancer's genetic mutation.

Investigators will do a kind of genetic testing called "DNA sequencing". Everyone who takes part in this trial will have genetic testing done on their cancer tumor tissue here at Dartmouth. The results of the DNA sequencing will be sent to N-of-One as noted above.

The treatment participants get will depend on the results of the DNA sequencing and the availability of targeted therapies that match the genetic profile of the tumor identified by the DNA sequencing.

If there is no genetic mutation that can be identified with current DNA sequencing, participants will receive the standard treatment for metastatic cancer.

If there is a genetic mutation that can be identified with current DNA sequencing and a drug has been developed for this mutation, participants may be able to receive that drug. If there is more than one drug available, the participant and his/her oncologist will decide which is the best one for the participant.

Because there are many drugs that may be used in this study, the investigator cannot advise in advance whether or not the drug a participant might receive has been approved by the U.S. Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Treatment with a personalized targeted therapy plan based on cancer genetics will improve time to disease progression (TTP) compared to standard therapies.

By comparing A) a patient's TTP on targeted therapy vs. B) their TTP on their most recent prior therapy, investigators will minimize the variability in TTP observed across cancer subtypes, and be able to enroll patients with any type of solid tumor in a statistically unbiased manner. Based on the literature, investigators expect at least 35% of patients treated with a genetically-informed targeted therapy to exhibit a longer progression-free interval than would be expected with standard therapies. This "TTP ratio" for each patient is calculated using the formula:

TTP ratio: (TTP on targeted therapy) / (TTP on most recent non-targeted therapy)

An individual patient's benefit from genetically-informed targeted therapy is defined as a TTP ratio ≥ 1.3

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic cancer that has progressed by RECIST criteria on at least 1 prior therapy in the metastatic setting.
* Patients must have not received anti-cancer therapy (i.e., EGFR, BRAF, AR, ER or Her2 targeted agents , chemotherapy, radiation or surgery) within the last 4 weeks, and must have recovered to Grade 2 or better from all treatment-related adverse events.
* Karnofsky performance status ≥ 60%
* Women should not be lactating or pregnant. If of childbearing age, she must have a negative pregnancy test within two weeks of entry to the study and practice effective birth control during the study.
* Patient must be mentally competent and provide written informed consent for study participation.
* Tumor tissue must be obtained through a clinically indicated biopsy or surgical procedure, performed as standard-of-care for progression of disease.
* Patient must consent to the use of blood, plasma, and tumor tissues for research purposes. Only tumor genetic information will be used to recommend therapy in this study. Tumor, blood and/ or plasma may be retrospectively analyzed for research purposes.
* Patients must be willing to consent to paying for the supply of drug if necessary. Cost estimates will be provided at the time of consent. As per the current standard of care for prescription drugs, the treating oncologist and his/her staff will be responsible for making every effort to obtain reimbursement and/or find the lowest possible cost of drug to minimize out of pocket costs.

Exclusion Criteria:

* Concomitant second invasive malignancy within five years of enrollment except for non- melanoma skin cancer.
* In patients with a prior history of invasive malignancy, less than five years in complete remission.
* Evidence of significant comorbidities such as uncontrolled diabetes, hypertension or active infection that would preclude treatment on a proposed regimen.
* Prior treatment with proposed regimen.
* Clinically significant gastrointestinal abnormalities including but not limited to malabsorption syndrome, major resection of stomach or small bowel affecting absorption of oral drugs, active peptic ulcer disease, inflammatory bowel disease, history of small bowel obstruction abscess or fistula within 28 days prior to beginning study treatment.
* Presence of uncontrolled infection.
* Known lesion infiltrating major vessels, with risk of bleeding or perforation, as determined by radiographic review.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.
* Any ongoing toxicity from prior anti-cancer therapy that is Grade 3 or higher and /or progressing in severity.
* Untreated brain metastasis that have progressed within the 8-week period prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | up to week 100
  All patients considered for entry should be consented and have measurable disease as described in the Response Evaluation Criteria in Solid Tumors criteria. Within 4 weeks of cycle 1 day 1 the following are required:
  * CT Chest/abdomen/pelvis with contrast and bone scan or PET scan
  * Brain MRI or CT head with contrast- if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States